CLINICAL TRIAL: NCT00251251
Title: Resynchronization/Defibrillation for Ambulatory Heart Failure Trial
Acronym: RAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Medtronic (Industry)
Responsible Party: Principal Investigator, Anthony Tang, Principal Investigator, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRN 63208; FRN 63208
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure, Congestive
Keywords: Congestive heart failure; Multicentre randomized controlled trial; Defibrillator; Cardiac resynchronization; Sudden death/mortality; Hospitalization; ICD indication; NYHA Class II; LVEF </equal to 30%; QRS >/equal to 120 ms
MeSH Terms: conditions — Heart Failure; Death, Sudden | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Optimal Medical therapy plus ICD (Active Comparator)
  Interventions: Device: Optimal Medical Therapy plus ICD
- 2. Optimal Medical Therapy plus CRT/ICD (Active Comparator)
  Interventions: Device: Optimal Medical Therapy plus CRT/ICD

INTERVENTIONS:
Device: Optimal Medical Therapy plus ICD — ICD vs CRT/ICD
  Arms: 1. Optimal Medical therapy plus ICD
Device: Optimal Medical Therapy plus CRT/ICD — ICD vs CRT/ICD
  Arms: 2. Optimal Medical Therapy plus CRT/ICD

SUMMARY:
Congestive heart failure (CHF) is a common health problem that leads to frequent hospitalizations and an increased death rate. In spite of advances in drug therapy, it remains a significant public health problem. Recently, a new therapy has been developed for advanced heart failure patients with a ventricular conduction abnormality. This new therapy, called cardiac resynchronization (CRT), is a device which stimulates the atrium, the right ventricle, and the left ventricle providing synchronization of the contraction of the heart chambers. It is the addition of this therapy to an implantable cardioverter defibrillator (ICD) that will be evaluated in this study. This study will compare whether the implantation of this new therapy device, in combination with an implantable cardioverter defibrillator, will reduce total mortality and hospitalizations for CHF.

DETAILED DESCRIPTION:
Cardiovascular mortality is decreasing in most industrial countries, however mortality for congestive heart failure is increasing. The most important predictors of mortality in heart failure patients are depressed left ventricular function, severity of symptoms (NYHA class), and ventricular conduction abnormality manifested as wide QRS. Recent advances in pharmacological therapy including ACE inhibitors, beta-blocker and spironolactone have resulted in improvement of symptoms and reduction in mortality. Population epidemiological studies demonstrated that mortality and hospitalization rate for heart failure remains very high despite recent pharmacological therapeutic progress. Recent short-term clinical trials demonstrated that cardiac resynchronization therapy (CRT) is effective in improving symptoms of heart failure, functional capacity and quality of life in patients with moderate to severe heart failure and conduction abnormality optimally treated with drug therapy. However, the data for morbidity and mortality in mild to moderate heart failure is lacking.

The objective of this trial is to determine if the addition of CRT to optimal pharmacological therapy and ICD is effect in reducing mortality and morbidity in patients with poor LV function, wide QRS and mild to moderate heart failure symptoms.

This is a double-blinded randomized control trial. A total of 1800 patients with mild to moderate heart failure symptoms, LVEF ≤ 30%, and QRS ≥ 120 ms will be included in the study. Patients will be randomized to either "ICD plus Optimal Medical Therapy (control)" or "CRT/ICD plus Optimal Medical Therapy (experimental)" in a 1:1 randomization ratio. Patients in the control group will be implanted with a single or dual chamber ICD. Patients in the experimental group will receive a device with the capabilities of CRT and ICD. Optimal Medical Therapy will include ACE inhibitors and beta-blockers. Patients will be followed on a regular basis and will have clinical evaluation, quality of life assessment, and six minute walk tests performed. The primary outcome is a composite of total mortality and heart failure hospitalization. Secondary outcome measures will include total mortality, cardiovascular mortality, sudden arrhythmic death, health related quality of life and cost economics. Patient accruement is scheduled for 4.5 years and a minimum follow of 18 months.

DFT sub study:

Overview of sub-study Design Patients participating in the RAFT trial, at participating sites, will be randomized to have DFT testing or no testing at the time of device implant. Up to 450 patients will be eligible for enrollment at Canadian and European centres. The study will have two primary outcomes: a short-term safety outcome and a long-term efficacy outcome. The safety outcome will be a composite of all adverse events potentially related to DFT that occur within 30 days following ICD implant. The long-term efficacy outcome will be a composite of failed first appropriate clinical ICD shock and sudden death. This pilot study is intended primarily to confirm the anticipated rates of events and to demonstrate feasibility of enrollment, but will not have statistical power to determine if intra-operative DFT testing is associated with significant short-term risk. If complication rates are as high as predicted and enrollment is feasible, then a larger study would be justified to determine the impact of intra-operative DFT testing on long-term rates of failed appropriated ICD shocks and sudden death. Events rates determined in this pilot study would then be used to estimate the sample size of this larger study.

Sub-study Long-Term Outcomes of the Resynchronization-Defibrillation for Ambulatory Heart Failure Trial (RAFT)

Coordinating Investigator:

John L. Sapp, Jr., MD, FRCPC

Funder:

John Sapp, QEII Div. of Cardiology, Halifax, NS

Coordinating Center:

QEII Heart Rhythm Research, Halifax, NS

The Resynchronization-Defibrillation for Ambulatory Heart Failure Trial (RAFT) was a multicenter, double-blind, randomized, controlled trial that aimed to determine whether the addition of CRT to an ICD, along with optimal medical therapy would reduce mortality and the rate of hospitalizations for HF, as compared to an ICD and optimal medical therapy alone. However, despite the established benefits of CRT among patients with mild to moderate HF, long term data is still lacking. We propose to determine the sustained, long-term outcomes of CRT among this high-risk patient population. A total of 8 sites enrolled more than 100 patients. Those 8 sites will ascertain long-term rates of survival, heart transplant and implantation of ventricular assist devices in a total of 1050 patients. The primary outcome will be all cause mortality. A secondary outcome will be the composite of mortality, implantation of ventricular assist device, and transplant. The 8 sites include UOHI, LHSC, QEII, Libin CV Calgary, HHSC, MHI, VCAT and Mazankowski Alberta Heart Institute.

The primary outcome is mortality (all cause). The primary analysis will compare the CRT-D and ICD groups for time to mortality. The survival experience (time-to-event) in each of the two groups will be analyzed using Kaplan-Meier product limit estimates and the nonparametric log-rank test. The hazard ratio (HR) and associated 95% CI will be calculated. In addition, the Cox proportional hazards model will be used to assess the consistency of the therapy group effect on this outcome taking the randomization stratification factors (clinical center, atrial rhythm (atrial fibrillation or flutter or sinus-atrial pacing), and a planned implantation of a single- or dual-chamber ICD)); as well, the Cox proportional hazards model analysis will be conducted as a sensitivity analysis to assess the therapy group effect on mortality while accounting for important baseline characteristics (any variable with a p value of less than 0.10 at baseline). Underlying assumptions for these statistical procedures will be assessed; in particular, the proportional hazard's assumption will be assessed using graphical (i.e., visual inspection of the log-negative-log plot) and numerical tests (i.e., test of the interaction term group x time). Should this assumption fail, a stratified Cox model will be fitted in order to correct for non-proportional hazards or, if ineffective, time-dependent variables will be introduced. In addition, chi-square tests will be used to compare the Kaplan-Meier (actuarial) rate of event-free survival at 10 years. The ITT population will be used.

The secondary outcome is the composite outcome of ventricular assist device implant (LVAD) or heart transplant or mortality (all cause). The primary analysis will compare the CRT-d and ICD groups for this composite outcome. For this analysis, the time-to-event analysis for Study Questions 1 will be followed. In addition, chi-square tests will be used to compare the Kaplan-Meier (actuarial) rate of event-free survival at 10 years. Also, the event rates for the composite outcome will be calculated for each therapy group and the relative risk (RR) and 95% CI calculated.

Secondary analysis - As a sensitivity analysis, the analysis for the primary and secondary questions 1 and will be repeated for the PP population.

Subgroup analysis - Subgroup analyses based on patient characteristics will be undertaken, primarily for sensitivity analyses to assess the robustness of the results, as well as for exploratory purposes for hypothesis generation. In particular, planned subgroups include: age (<65, ≥65), sex (male, female), NYHA Class (I, II), ischemic heart disease (<150, ≥150) paced QRS, LV ejection fraction, atrial rhythm (permanent Afib/flutter, sinus or atrial paced). The interaction of the therapy and subgroup will be included in the models.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) Class II
* Left ventricular ejection fraction (LVEF) less than or equal to 30% by multigated acquisition scan (MUGA)/catheterization OR LVEF less than or equal to 30% and LV end diastolic dimension ≥ 60 mm (by echocardiogram) within 6 months prior to randomization
* Intrinsic QRS complex width ≥ 120 ms OR paced QRS measurement ≥ 200 ms
* ICD indication for primary or secondary prevention
* Optimal heart failure pharmacological therapy
* Normal sinus rhythm; OR chronic persistent atrial tachyarrhythmia with resting ventricular heart rate ≤ 60 beats per minute (bpm) and 6 minute hall walk ventricular heart rate of ≤ 90 bpm; OR chronic persistent atrial tachyarrhythmia with resting ventricular heart rate > 60 bpm and 6 minute hall walk ventricular heart rate of > 90 bpm and booked for atrioventricular junction ablation.

Exclusion Criteria:

* Intravenous inotropic agent in the last 4 days
* Patients with a life expectancy of less than one year from non-cardiac cause
* Expected to undergo cardiac transplantation within one year (status I)
* In hospital patients who have acute cardiac or non-cardiac illness that requires intensive care
* Uncorrected or uncorrectable primary valvular disease
* Restrictive, hypertrophic, or reversible form of cardiomyopathy
* Severe primary pulmonary disease such as cor pulmonale
* Tricuspid prosthetic valve
* Patients with an existing ICD (patients with an existing pacemaker may be included if the patients satisfy all other inclusion/exclusion criteria)
* Coronary revascularization (coronary artery bypass graft surgery [CABG] or percutaneous coronary intervention [PCI]) < 1 month if previously determined LVEF > 30%. Patients with a more recent revascularization can be included if a previously determined LVEF was ≤ 30%.
* Patients with an acute coronary syndrome including myocardial infarction (MI) can be included if the patients have had a previous MI with LV dysfunction (LVEF ≤ 30%).
* Patients included in another clinical trial that will affect the objectives of this study
* History of noncompliance to medical therapy
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1798 (Actual)
Dates: Start 2003-04; Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Primary outcome is a composite of all cause total mortality and hospitalization for CHF | Study end

SECONDARY OUTCOMES:
Total mortality | Study end
Cardiovascular mortality | Study end
Sudden arrhythmic death | Study end
Progressive HF death | Study end
All cause hospitalization rate | Study end
CHF hospitalization rate | Study end
Health related quality of life | Study end
Cost economics | Study end

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Tang, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; George Wells, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (33):
- Australia (2):
  - Royal Adelaide Hospital, Adelaide
  - Sir Charles Gairdner Hospital, Perth
- University Ziekenhuis, Leuven, Belgium
- Canada (22):
  - University of Calgary/Foothill Hospital, Calgary, Alberta
  - Alberta Heart Institute, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - NB Heart Centre Research Initiative, Saint John, New Brunswick
  - Memorial Hospital, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - St. Mary's Hospital, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Care, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - UHN Toronto General, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM Hopital Notre Dame, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hopital du Sacre Coeur de Montreal, Montreal, Quebec
  - Laval Hospital, Québec, Quebec
  - CHUS Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Skejby University Hospital, Aarhus, Denmark
- Germany (5):
  - Zentralklinik, Bad Berka
  - J.W. Goethe University, Frankfurt
  - University of Giessen, Giessen
  - Ludwigshafen, Ludwigshafen
  - University of Mainz, Mainz
- Isala Klinieken, Zwolle, Netherlands
- Ege University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Sapp JL, Sivakumaran S, Redpath CJ, Khan H, Parkash R, Exner DV, Healey JS, Thibault B, Sterns LD, Lam NHN, Manlucu J, Mokhtar A, Sumner G, McKinlay S, Kimber S, Mondesert B, Talajic M, Rouleau J, McCarron CE, Wells G, Tang ASL; RAFT Long-Term Study Team. Long-Term Outcomes of Resynchronization-Defibrillation for Heart Failure. N Engl J Med. 2024 Jan 18;390(3):212-220. doi: 10.1056/NEJMoa2304542. PMID 38231622
- [Derived] Fudim M, Dalgaard F, Friedman DJ, Abraham WT, Cleland JGF, Curtis AB, Gold MR, Kutyifa V, Linde C, Ali-Ahmed F, Tang A, Olivas-Martinez A, Inoue LYT, Al-Khatib SM, Sanders GD. Comorbidities and clinical response to cardiac resynchronization therapy: Patient-level meta-analysis from eight clinical trials. Eur J Heart Fail. 2024 Apr;26(4):1039-1046. doi: 10.1002/ejhf.3029. Epub 2023 Sep 15. PMID 37671601
- [Derived] Friedman DJ, Al-Khatib SM, Dalgaard F, Fudim M, Abraham WT, Cleland JGF, Curtis AB, Gold MR, Kutyifa V, Linde C, Tang AS, Ali-Ahmed F, Olivas-Martinez A, Inoue LYT, Sanders GD. Cardiac Resynchronization Therapy Improves Outcomes in Patients With Intraventricular Conduction Delay But Not Right Bundle Branch Block: A Patient-Level Meta-Analysis of Randomized Controlled Trials. Circulation. 2023 Mar 7;147(10):812-823. doi: 10.1161/CIRCULATIONAHA.122.062124. Epub 2023 Jan 26. PMID 36700426
- [Derived] Manlucu J, Sharma V, Koehler J, Warman EN, Wells GA, Gula LJ, Yee R, Tang AS. Incremental Value of Implantable Cardiac Device Diagnostic Variables Over Clinical Parameters to Predict Mortality in Patients With Mild to Moderate Heart Failure. J Am Heart Assoc. 2019 Jul 16;8(14):e010998. doi: 10.1161/JAHA.118.010998. Epub 2019 Jul 11. PMID 31291801
- [Derived] Bennett MT, Leader N, Sapp J, Parkash R, Gardner M, Healey JS, Thibault B, Sterns L, Essebag V, Birnie D, Sivakumaran S, Nery P, Andrade JG, Krahn AD, Tang A. Differentiating Ventricular From Supraventricular Arrhythmias Using the Postpacing Interval After Failed Antitachycardia Pacing. Circ Arrhythm Electrophysiol. 2018 Apr;11(4):e005921. doi: 10.1161/CIRCEP.117.005921. PMID 29618476
- [Derived] Linde C, Cleland JGF, Gold MR, Claude Daubert J, Tang ASL, Young JB, Sherfesee L, Abraham WT. The interaction of sex, height, and QRS duration on the effects of cardiac resynchronization therapy on morbidity and mortality: an individual-patient data meta-analysis. Eur J Heart Fail. 2018 Apr;20(4):780-791. doi: 10.1002/ejhf.1133. Epub 2018 Jan 4. PMID 29314424
- [Derived] Sapp JL, Parkash R, Wells GA, Yetisir E, Gardner MJ, Healey JS, Thibault B, Sterns LD, Birnie D, Nery PB, Sivakumaran S, Essebag V, Dorian P, Tang AS. Cardiac Resynchronization Therapy Reduces Ventricular Arrhythmias in Primary but Not Secondary Prophylactic Implantable Cardioverter Defibrillator Patients: Insight From the Resynchronization in Ambulatory Heart Failure Trial. Circ Arrhythm Electrophysiol. 2017 Mar;10(3):e004875. doi: 10.1161/CIRCEP.116.004875. PMID 28292754
- [Derived] Wilton SB, Exner DV, Wyse DG, Yetisir E, Wells G, Tang AS, Healey JS. Frequency and Outcomes of Postrandomization Atrial Tachyarrhythmias in the Resynchronization/Defibrillation in Ambulatory Heart Failure Trial. Circ Arrhythm Electrophysiol. 2016 May;9(5):e003807. doi: 10.1161/CIRCEP.115.003807. PMID 27162033
- [Derived] Gillis AM, Kerr CR, Philippon F, Newton G, Talajic M, Froeschl M, Froeschl S, Swiggum E, Yetisir E, Wells GA, Tang AS. Impact of cardiac resynchronization therapy on hospitalizations in the Resynchronization-Defibrillation for Ambulatory Heart Failure trial. Circulation. 2014 May 20;129(20):2021-30. doi: 10.1161/CIRCULATIONAHA.112.000417. Epub 2014 Mar 7. PMID 24610807
- [Derived] Birnie DH, Ha A, Higginson L, Sidhu K, Green M, Philippon F, Thibault B, Wells G, Tang A. Impact of QRS morphology and duration on outcomes after cardiac resynchronization therapy: Results from the Resynchronization-Defibrillation for Ambulatory Heart Failure Trial (RAFT). Circ Heart Fail. 2013 Nov;6(6):1190-8. doi: 10.1161/CIRCHEARTFAILURE.113.000380. Epub 2013 Aug 30. PMID 23995437
- [Derived] Cleland JG, Abraham WT, Linde C, Gold MR, Young JB, Claude Daubert J, Sherfesee L, Wells GA, Tang AS. An individual patient meta-analysis of five randomized trials assessing the effects of cardiac resynchronization therapy on morbidity and mortality in patients with symptomatic heart failure. Eur Heart J. 2013 Dec;34(46):3547-56. doi: 10.1093/eurheartj/eht290. Epub 2013 Jul 29. PMID 23900696
- [Derived] Healey JS, Hohnloser SH, Exner DV, Birnie DH, Parkash R, Connolly SJ, Krahn AD, Simpson CS, Thibault B, Basta M, Philippon F, Dorian P, Nair GM, Sivakumaran S, Yetisir E, Wells GA, Tang AS; RAFT Investigators. Cardiac resynchronization therapy in patients with permanent atrial fibrillation: results from the Resynchronization for Ambulatory Heart Failure Trial (RAFT). Circ Heart Fail. 2012 Sep 1;5(5):566-70. doi: 10.1161/CIRCHEARTFAILURE.112.968867. Epub 2012 Aug 14. PMID 22896584
- [Derived] Healey JS, Gula LJ, Birnie DH, Sterns L, Connolly SJ, Sapp J, Crystal E, Simpson C, Exner DV, Kus T, Philippon F, Wells G, Tang AS. A randomized-controlled pilot study comparing ICD implantation with and without intraoperative defibrillation testing in patients with heart failure and severe left ventricular dysfunction: a substudy of the RAFT trial. J Cardiovasc Electrophysiol. 2012 Dec;23(12):1313-6. doi: 10.1111/j.1540-8167.2012.02393.x. Epub 2012 Jul 12. PMID 22788915
- [Derived] Tang AS, Wells GA, Talajic M, Arnold MO, Sheldon R, Connolly S, Hohnloser SH, Nichol G, Birnie DH, Sapp JL, Yee R, Healey JS, Rouleau JL; Resynchronization-Defibrillation for Ambulatory Heart Failure Trial Investigators. Cardiac-resynchronization therapy for mild-to-moderate heart failure. N Engl J Med. 2010 Dec 16;363(25):2385-95. doi: 10.1056/NEJMoa1009540. Epub 2010 Nov 14. PMID 21073365